CLINICAL TRIAL: NCT06667713
Title: ENTRUST - Economic Navigation and Strengthening to Realize Unrestricted Services for Transgender Women
Acronym: ENTRUST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped because of executive orders of new administration
Sponsor: University of Central Florida (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elena Cyrus, Associate Professor of Medicine, University of Central Florida
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: University of Central Florida; DP2DA058436 (NIH)
Record Dates: First submitted 2024-10-21; First posted 2024-10-31 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Substance Use Disorder (SUD); HIV
Keywords: economic strengthening; substance use; HIV; Florida
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): ENTRUST intervention comprised of adapted SBIRT-T, economic strengthening and photovoice training
  Interventions: Behavioral: ENTRUST - substance use and HIV counseling and goal setting with economic empowerment and photovoice training
- Waitlist Control (Active Comparator): SBIRT-T only
  Interventions: Behavioral: SBIRT-T only

INTERVENTIONS:
Behavioral: ENTRUST - substance use and HIV counseling and goal setting with economic empowerment and photovoice training — The ENTRUST intervention consists of an adapted counseling intervention based on motivational interviewing techniques and goal setting (SBIRT-T); Economic skill building using a tailored app (WorthIt for ENTRUST); and, Photovoice Activities with an optional photo exhibit
  Arms: Intervention
Behavioral: SBIRT-T only — An adapted screening brief intervention and referral to treatment intervention to link transgender women to substance use and HIV services
  Arms: Waitlist Control

SUMMARY:
Transgender women in Florida are economically disadvantaged and at highest risk for substance use disorders, HIV transmission and/or non-adherence to antiretroviral treatment, yet remain underrepresented in research. Existing programs fail to address structural barriers such as socio-economic status and social marginalization that deter access to prevention services and care. For this study, acceptability, feasibility, and preliminary efficacy of ENTRUST (economic navigation and strengthening to realize unrestricted services for transgender women) will be assessed. ENTRUST is an economic-based empowerment intervention that will provide transgender women with group-based financial education while receiving tailored SBIRT counseling to help transgender women routinely engaging in substance use services and HIV care or preexposure prophylaxis (PrEP) programs. Participants will be assigned to either the ENTRUST intervention arm or a waitlist control arm. Participants in the intervention arm will receive the ENTRUST intervention during 6-month follow up, and participants assigned to the control arm will have the option of receiving the ENTRUST intervention at the end of the study. Participants in the intervention arm must complete about half of the visits in person, and participants in the control arm will have the option of completing the study visits remotely or in person. All participants will be followed for six months and will complete 4 - 15 study visits. In person site visits will occur at one of our participating sites in Orlando or Miami and will be conducted in English and/or Spanish only. Participants must be adults (over the age) and residing in South or Central Florida. Participants can be enrolled in the study for 6 - 8 months.

DETAILED DESCRIPTION:
The ENTRUST intervention is adaptive based on participant's substance use, HIV status and economic status. Participants in both arms will receive an adapted tailored screening, brief intervention and referral to treatment intervention for transgender women (SBIRT-T) to set personal goals around linking to substance use services, HIV care and linking to financial institutions. As indicated participants may also receive support with mental health services, housing and legal services. Any participant who receives the ENTRUST intervention will also participate in group-based economic empowerment and skill building training, and photovoice training. Photovoice is a process where participants take pictures of their daily lives while they are in the study to help document their experience. The economic empowerment training will be completed using a tailored app developed by the Human Rights Campaign for this Study (WorthIt for ENTRUST) over four sessions. The photovoice training will be facilitated by an ENTRUST facilitator at one of the participating collaborating sites in Orlando or Miami. At the end of the four photovoice sessions, participants may volunteer to do a public exhibit presenting study images from the photovoice activities to key stakeholders to initiate a call to action around policy to impact change that improves transgender women linking to substance use services and HIV care and improving their financial health.

ELIGIBILITY:
Inclusion Criteria:

Economically vulnerable adult transgender women at risk for SUD and/or HIV who speak English or Spanish and live in South or Central Florida

Exclusion Criteria:

Minor transgender women who do not speak English or Spanish and can not attend visits in South or Central Florida

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women assigned male at birth
Enrollment: 12 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Number of people engaging and being retained in substance use and HIV services | 6 months
  Engagement will be measured by self-report of at least one visit to a substance use treatment center/[HIV] provider during 6 month follow up A participant will be considered retained in care if they complete more than one treatment to the facility during 6 month follow up The number of visits will be reported for each facility by outcome (substance use or HIV prevention/treatment)
Number of people linking to other support services other than substance use or HIV services | 6 months
  Engagement will be measured by self-report of at least one visit to a bank or other similar financial entity/mental health/housing/legal service during 6 month follow up A participant will be considered retained in care if they complete more than one treatment to a facility during 6 month follow up The number of visits will be reported for each facility by outcome

SECONDARY OUTCOMES:
Substance Use Disorder Diagnosis | Any time during 6 months of follow up
  Per AUDIT and DAST criteria. Higher scores indicate a greater risk of developing an alcohol use (AUDIT) or drug use (DAST) disorder
HIV diagnosis | Any time during 6 months of follow up
  Measure by rapid oral swab and confirmed by Western Blot Confirmatory test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the sensitivity of the information that may deidentify participants, some variables may not be shared. However, there will be a plan to share deidentified data related to primary and secondary outcomes.

REFERENCES:
- [Background] Thoele K, Moffat L, Konicek S, Lam-Chi M, Newkirk E, Fulton J, Newhouse R. Strategies to promote the implementation of Screening, Brief Intervention, and Referral to Treatment (SBIRT) in healthcare settings: a scoping review. Subst Abuse Treat Prev Policy. 2021 May 11;16(1):42. doi: 10.1186/s13011-021-00380-z. PMID 33975614
- [Background] Bray JW, Del Boca FK, McRee BG, Hayashi SW, Babor TF. Screening, Brief Intervention and Referral to Treatment (SBIRT): rationale, program overview and cross-site evaluation. Addiction. 2017 Feb;112 Suppl 2:3-11. doi: 10.1111/add.13676. PMID 28074566
- [Background] Singh M, Gmyrek A, Hernandez A, Damon D, Hayashi S. Sustaining Screening, Brief Intervention and Referral to Treatment (SBIRT) services in health-care settings. Addiction. 2017 Feb;112 Suppl 2:92-100. doi: 10.1111/add.13654. PMID 28074565
- [Background] Cyrus E, Johnson SA, Perez-Gilbe HR, Wuyke G, Fajardo FJ, Garba NA, Devieux J, Jimenez D, Garcia S, Holder CL. Engagement in Care and Housing Instability Influence HIV Screening Among Transgender Individuals in South Florida. Transgend Health. 2022 Feb 14;7(1):52-60. doi: 10.1089/trgh.2020.0066. eCollection 2022 Feb. PMID 35224190
- [Background] Holder CL, Perez-Gilbe HR, Fajardo FJ, Garcia S, Cyrus E. Disparities of HIV risk and PrEP use among transgender women of color in South Florida. J Natl Med Assoc. 2019 Dec;111(6):625-632. doi: 10.1016/j.jnma.2019.08.001. Epub 2019 Sep 13. PMID 31526532
- See also: Link to adapted HRC app for ENTRUST economic strengthening — https://worthitforentrust.hrc.org/